CLINICAL TRIAL: NCT03580434
Title: National, Multicentre, Pilot Study, to Evaluate Safety and Performance of the V-STRUT© Transpedicular Vertebral System Indicated for Vertebral Compression Fracture Treatment
Brief Title: The Purpose of This Study is to Evaluate Safety and Performance of the V-STRUT© Transpedicular Vertebral System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyprevention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPINE0
Record Dates: First submitted 2018-06-04; First posted 2018-07-09 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Vertebral Compression Fracture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-STRUT (Experimental): V-STRUT implantation
  Interventions: Device: V-STRUT

INTERVENTIONS:
Device: V-STRUT — Minimally invasive implantation of V-STRUT

SUMMARY:
The purpose of this pilot study is to evaluate the safety and performance of the V-STRUT© Transpedicular Vertebral System for the treatment of vertebral compression fractures of the thoracic or lumbar spine.

ELIGIBILITY:
Inclusion Criteria :

* Adult male and female patients
* Treatment of vertebral compression fracture (type A.1, some A.2 and rarely A.3 Magerl classification)
* Due to osteoporosis or tumorous lesions,
* Located in the thoracic and/or lumbar spine from T9 to L5.
* One unique vertebral fracture to be treated with the device
* Pain > 4
* ASA > 5
* For osteoporotic patient, fail in conservative treatment (8 days of antalgic medication Level III) and recent fracture (less than 6 weeks).

Exclusion Criteria:

* Unstable fractures or neoplasms with posterior involvement
* Nonmobile fractures
* Damages of the pedicles or posterior wall
* Less than one third of the original vertebral body height remaining
* Spinal canal stenosis (>20%)
* Neurologic signs or symptoms related to the compression fracture or impeding pathological fracture
* Patient clearly improving on conservative treatment
* Pregnancy, breastfeeding
* Any contra-indication / allergy to implant material or cement
* Any previous surgical treatment (material or cement) in the targeted vertebra
* Systemic infection or infection located in the spine
* Any medical condition including but not limited to anaemia, coagulation disorders, fibromyalgia, algoneurodystrophy, Paget's disease, uncontrolled diabetes that would preclude the patient from having surgery or would impede the benefit of surgery
* Patient under the age of majority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Difficulties of the procedure [feasibility of the procedure] | per-operative
  Record difficulties experienced by surgeons during the procedure: each individual step of the procedure will be recorded and quoted by practitioners as very easy, easy, difficult or very difficult.
Type of anaesthesia [feasibility of the procedure] | per-operative
  Record the type of anaesthesia as GA (General Anaesthesia), local anaesthesia + sedation, or other.
Cement quantity injected [feasibility of the procedure] | per-operative
  Record cement quantity injected in the vertebral body, in cc (cubic centimeter).
Operating time [feasibility of the procedure] | per-operative
  Measuring the duration of the surgical procedures.
Hospitalisation stay [feasibility of the procedure] | per-operative and immediate post-op
  Measuring the duration of the hospitalisation stay.

SECONDARY OUTCOMES:
Pain [performance of the device] | pre- operative, immediate post-op, at 2 months, 6 months and 12 months.
  Self-evaluation of pain using Visual Analogue Scale (VAS) going from 0 (no pain) to 10 (maximum).
Frequencies of ADEs and SADEs [safety of the device] | per- operative, immediate post-op, at 2 months, 6 months and 12 months.
  Measuring the frequencies of Adverse Device-related Events (ADEs) and Severe Adverse Device-related Events (SADEs).
Rates of cement leakage [safety of the device] | Per-operative, immediate post-op, at 2 months, 6 months and 12 months.
  Measuring the rates of cement leakages.
Rates of fractures [safety of the device] | Per-operative, immediate post-op, at 2 months, 6 months and 12 months.
  Measuring the rates of subsequent, adjacent and pedicle fractures.
Functional score [safety of the device] | per-operative, immediate post-op, at 2 months, 6 months and 12 months.
  Measuring patient's disability using the 100 points ODI (Oswestry Disability Index) functional score.
Haematomas and infections rates [safety of the device] | per-operative, immediate post-op, at 2 months, 6 months and 12 months.
  Measuring haematomas and infections rates.
Wound healing [safety of the device] | per-operative, immediate post-op, at 2 months, 6 months and 12 months.
  Assessment of wound-healing by practitioners.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - APHP - Hôpital Tenon, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The data analysis of the investigation will carry out a final report that will be sent to the CPP and ANSM.
  According to the law N°2002-303 dated March 4, 2002, the patients involved in the study will be informed on demand on the global data analysis.
  Regarding publication, if the data analysis provides important and interesting information on the device and its associated procedure for the treatment of vertebral compression fracture which aims to complete the state of the art, it may be decided to publish the corresponding data. In this case, the IPD that will be shared will consists of all IPD that underlie results in this publication.

REFERENCES:
- [Background] Cornelis FH, Tselikas L, Carteret T, Lapuyade B, De Baere T, Le Huec JC, Deschamps F. Percutaneous internal fixation with Y-STRUT(R) device to prevent both osteoporotic and pathological hip fractures: a prospective pilot study. J Orthop Surg Res. 2017 Feb 9;12(1):27. doi: 10.1186/s13018-017-0514-2. PMID 28183325
- [Background] Cornelis FH, Deschamps F. Augmented osteoplasty for proximal femur consolidation in cancer patients: Biomechanical considerations and techniques. Diagn Interv Imaging. 2017 Sep;98(9):645-650. doi: 10.1016/j.diii.2017.06.014. Epub 2017 Jul 27. PMID 28757428
- [Background] Cornelis FH, Tselikas L, Carteret T, Lapuyade B, De Baere T, Cabane V, Rodrigues L, Maas C, Deschamps F. A Novel Implant for the Prophylactic Treatment of Impending Pathological Fractures of the Proximal Femur: Results from a Prospective, First-in-Man Study. Cardiovasc Intervent Radiol. 2017 Jul;40(7):1070-1076. doi: 10.1007/s00270-017-1613-5. Epub 2017 Feb 23. PMID 28233056
- [Background] Szpalski M,Le Huec JC, Jayankura M, Reynders P, Maas C(2017) Contralateral Prophylactic Reinforcement in Case of First Low-Energy Hip Fracture: First-in-Man Clinical Data of a New Percutaneous Internal Fixation Device. J Osteopor Phys Act 5:202. doi:10.4172/2329-9509.100020
- [Background] Upasani VV, Robertson C, Lee D, Tomlinson T, Mahar AT. Biomechanical comparison of kyphoplasty versus a titanium mesh implant with cement for stabilization of vertebral compression fractures. Spine (Phila Pa 1976). 2010 Sep 1;35(19):1783-8. doi: 10.1097/BRS.0b013e3181b7cc5d. PMID 20098352
- [Background] Ghofrani H, Nunn T, Robertson C, Mahar A, Lee Y, Garfin S. An evaluation of fracture stabilization comparing kyphoplasty and titanium mesh repair techniques for vertebral compression fractures: is bone cement necessary? Spine (Phila Pa 1976). 2010 Jul 15;35(16):E768-73. doi: 10.1097/BRS.0b013e3181d260bf. PMID 20634659
- [Background] Belkoff SM, Mathis JM, Jasper LE. Ex vivo biomechanical comparison of hydroxyapatite and polymethylmethacrylate cements for use with vertebroplasty. AJNR Am J Neuroradiol. 2002 Nov-Dec;23(10):1647-51. PMID 12427616
- [Background] Rodrigues DC, Ordway NR, Ma CR, Fayyazi AH, Hasenwinkel JM. An ex vivo exothermal and mechanical evaluation of two-solution bone cements in vertebroplasty. Spine J. 2011 May;11(5):432-9. doi: 10.1016/j.spinee.2011.02.012. Epub 2011 Apr 11. PMID 21481652
- [Background] Tutton SM, Pflugmacher R, Davidian M, Beall DP, Facchini FR, Garfin SR. KAST Study: The Kiva System As a Vertebral Augmentation Treatment-A Safety and Effectiveness Trial: A Randomized, Noninferiority Trial Comparing the Kiva System With Balloon Kyphoplasty in Treatment of Osteoporotic Vertebral Compression Fractures. Spine (Phila Pa 1976). 2015 Jun 15;40(12):865-75. doi: 10.1097/BRS.0000000000000906. PMID 25822543
- [Background] Dohm M, Black CM, Dacre A, Tillman JB, Fueredi G; KAVIAR investigators. A randomized trial comparing balloon kyphoplasty and vertebroplasty for vertebral compression fractures due to osteoporosis. AJNR Am J Neuroradiol. 2014 Dec;35(12):2227-36. doi: 10.3174/ajnr.A4127. Epub 2014 Oct 9. PMID 25300981
- [Background] Olivarez LM, Dipp JM, Escamilla RF, Bajares G, Perez A, Stubbs HA, Block JE. Vertebral augmentation treatment of painful osteoporotic compression fractures with the Kiva VCF Treatment System. SAS J. 2011 Dec 1;5(4):114-9. doi: 10.1016/j.esas.2011.06.001. eCollection 2011. PMID 25802677
- [Background] Wang CH, Ma JZ, Zhang CC, Nie L. Comparison of high-viscosity cement vertebroplasty and balloon kyphoplasty for the treatment of osteoporotic vertebral compression fractures. Pain Physician. 2015 Mar-Apr;18(2):E187-94. PMID 25794218
- [Background] Li X, Yang H, Tang T, Qian Z, Chen L, Zhang Z. Comparison of kyphoplasty and vertebroplasty for treatment of painful osteoporotic vertebral compression fractures: twelve-month follow-up in a prospective nonrandomized comparative study. J Spinal Disord Tech. 2012 May;25(3):142-9. doi: 10.1097/BSD.0b013e318213c113. PMID 21423053
- [Background] Deschamps F, de Baere T. Cementoplasty of bone metastases. Diagn Interv Imaging. 2012 Sep;93(9):685-689. doi: 10.1016/j.diii.2012.06.009. Epub 2012 Aug 11. PMID 22889809
- [Background] Kobayashi N, Numaguchi Y, Fuwa S, Uemura A, Matsusako M, Okajima Y, Ishiyama M, Takahashi O. Prophylactic vertebroplasty: cement injection into non-fractured vertebral bodies during percutaneous vertebroplasty. Acad Radiol. 2009 Feb;16(2):136-43. doi: 10.1016/j.acra.2008.05.005. PMID 19124098
- [Background] Otten LA, Bornemnn R, Jansen TR, Kabir K, Pennekamp PH, Wirtz DC, Stuwe B, Pflugmacher R. Comparison of balloon kyphoplasty with the new Kiva(R) VCF system for the treatment of vertebral compression fractures. Pain Physician. 2013 Sep-Oct;16(5):E505-12. PMID 24077200
- [Background] Yang EZ, Xu JG, Huang GZ, Xiao WZ, Liu XK, Zeng BF, Lian XF. Percutaneous Vertebroplasty Versus Conservative Treatment in Aged Patients With Acute Osteoporotic Vertebral Compression Fractures: A Prospective Randomized Controlled Clinical Study. Spine (Phila Pa 1976). 2016 Apr;41(8):653-60. doi: 10.1097/BRS.0000000000001298. PMID 26630417
- [Background] Korovessis P, Vardakastanis K, Repantis T, Vitsas V. Balloon kyphoplasty versus KIVA vertebral augmentation--comparison of 2 techniques for osteoporotic vertebral body fractures: a prospective randomized study. Spine (Phila Pa 1976). 2013 Feb 15;38(4):292-9. doi: 10.1097/BRS.0b013e31826b3aef. PMID 23407406
- [Background] Shindle MK, Gardner MJ, Koob J, Bukata S, Cabin JA, Lane JM. Vertebral height restoration in osteoporotic compression fractures: kyphoplasty balloon tamp is superior to postural correction alone. Osteoporos Int. 2006 Dec;17(12):1815-9. doi: 10.1007/s00198-006-0195-x. Epub 2006 Sep 16. PMID 16983458
- [Background] Liu JT, Li CS, Chang CS, Liao WJ. Long-term follow-up study of osteoporotic vertebral compression fracture treated using balloon kyphoplasty and vertebroplasty. J Neurosurg Spine. 2015 Jul;23(1):94-8. doi: 10.3171/2014.11.SPINE14579. Epub 2015 Apr 17. PMID 25884343
- [Background] Evans AJ, Kip KE, Brinjikji W, Layton KF, Jensen ML, Gaughen JR, Kallmes DF. Randomized controlled trial of vertebroplasty versus kyphoplasty in the treatment of vertebral compression fractures. J Neurointerv Surg. 2016 Jul;8(7):756-63. doi: 10.1136/neurintsurg-2015-011811. Epub 2015 Jun 24. PMID 26109687
- [Background] Chen D, An ZQ, Song S, Tang JF, Qin H. Percutaneous vertebroplasty compared with conservative treatment in patients with chronic painful osteoporotic spinal fractures. J Clin Neurosci. 2014 Mar;21(3):473-7. doi: 10.1016/j.jocn.2013.05.017. Epub 2013 Aug 8. PMID 24315046
- [Background] Comstock BA, Sitlani CM, Jarvik JG, Heagerty PJ, Turner JA, Kallmes DF. Investigational vertebroplasty safety and efficacy trial (INVEST): patient-reported outcomes through 1 year. Radiology. 2013 Oct;269(1):224-31. doi: 10.1148/radiol.13120821. Epub 2013 May 21. PMID 23696683
- [Background] Tan HY, Wang LM, Zhao L, Liu YL, Song RP. A prospective study of percutaneous vertebroplasty for chronic painful osteoporotic vertebral compression fracture. Pain Res Manag. 2015 Jan-Feb;20(1):e8-e11. doi: 10.1155/2015/181487. Epub 2014 Jun 19. PMID 24945287
- [Background] Korovessis P, Repantis T, Miller LE, Block JE. Initial clinical experience with a novel vertebral augmentation system for treatment of symptomatic vertebral compression fractures: a case series of 26 consecutive patients. BMC Musculoskelet Disord. 2011 Sep 22;12:206. doi: 10.1186/1471-2474-12-206. PMID 21939548
- [Background] Yi X, Lu H, Tian F, Wang Y, Li C, Liu H, Liu X, Li H. Recompression in new levels after percutaneous vertebroplasty and kyphoplasty compared with conservative treatment. Arch Orthop Trauma Surg. 2014 Jan;134(1):21-30. doi: 10.1007/s00402-013-1886-3. Epub 2013 Nov 28. PMID 24287674
- [Background] Vogl TJ, Pflugmacher R, Hierholzer J, Stender G, Gounis M, Wakhloo A, Fiebig C, Hammerstingl R. Cement directed kyphoplasty reduces cement leakage as compared with vertebroplasty: results of a controlled, randomized trial. Spine (Phila Pa 1976). 2013 Sep 15;38(20):1730-6. doi: 10.1097/BRS.0b013e3182a14d15. PMID 23804157